CLINICAL TRIAL: NCT02024178
Title: A Pilot Evaluation of the Efficacy of HistoScanning™ in Predicting the Presence and Location of Prostate Cancer in Men Undergoing Radical Prostatectomy
Brief Title: Ultrasound Imaging in Finding Prostate Cancer in Patients Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NYU11-00220
Record Dates: First submitted 2013-12-26; First posted 2013-12-31 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radical Prostatectomy; Ultrasound Imaging
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound Imaging (Experimental): Men already electing to undergo radical prostatectomy will undergo transrectal ultrasound procedure at induction of anesthesia prior to their surgery procedure.
  Interventions: Procedure: Ultrasound Imaging

INTERVENTIONS:
Procedure: Ultrasound Imaging

SUMMARY:
This pilot clinical trial studies ultrasound imaging in finding prostate cancer in patients undergoing surgery. Diagnostic procedures, such as ultrasound imaging, may help find and diagnose prostate cancer. This study will serve as an analysis of the Histo-Scanning technology for the purpose of determining its ability to identify sites of prostate cancer at the time of prostate ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed a staging multiparametric MRI at New York University (NYU)
* Patients who plan to undergo radical prostatectomy by open or robotic approach

Exclusion Criteria:

* Previous History of Prostate Cancer Radiation Treatment
* Focal Ablation of the prostate for cancer treatment
* Men receiving hormonal ablation within 6 months prior to undergoing radical prostatectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Correlation of Histoscan findings with Radical Prostatectomy Pathology | up to 3 years
  Compare location and concordance of findings on pre-op MRI & Histoscan with radical prostatectomy specimen

SECONDARY OUTCOMES:
Extent of tumor and grade in treatment planning | Up to 3 years
  Describe correlation between tumor grade on final pathology and histoscan findings

CONTACTS AND LOCATIONS:
Overall Officials: Samir Taneja, MD, Principal Investigator — NYU Langone Health
Locations (1):
- Smilow Comprehensive Prostate Cancer Center, New York, New York, United States